CLINICAL TRIAL: NCT02517684
Title: Top-down Infliximab Study in Kids With Crohn's Disease
Acronym: TISKids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Lissy de Ridder, Pediatric Gastroenterologist, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL52030.078.15; 2014-005702-37 (EudraCT Number); MEC-2015-080 (Other: Medical Ethical Trial Committee Erasmus MC)
Record Dates: First submitted 2015-07-01; First posted 2015-08-07 (Estimated); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; pediatric; infliximab; top-down; TISKids
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab; Prednisolone; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Top-down (Experimental): Infliximab and azathioprine; patients will receive 5 infliximab infusions of 5 mg/kg (IFX induction at week 0, 2 and 6, followed by 2 maintenance infusions every 8 weeks). IFX will be discontinued after 5 IFX infusions. Patients will also receive oral azathioprine 2-3 mg/kg, once daily as maintenance treatment.
  Interventions: Drug: Infliximab; Drug: Azathioprine
- Step-up (Active Comparator): Step-up treatment will consist of standard induction treatment by either oral prednisolone 1 mg/kg (maximum 40 mg) once daily for 4 weeks, followed by tapering in 6 weeks until stop, or EEN with polymeric feeding for 6-8 weeks after which normal foods are gradually reintroduced within 2-3 weeks. Either of these induction treatments will be combined with oral AZA 2-3 mg, once daily, as maintenance treatment.
  Interventions: Drug: Prednisolone; Other: Exclusive enteral nutrition; Drug: Azathioprine

INTERVENTIONS:
Drug: Infliximab
  Other Names: Inflectra
  Arms: Top-down
Drug: Prednisolone
  Arms: Step-up
Other: Exclusive enteral nutrition
  Arms: Step-up
Drug: Azathioprine
  Other Names: Imuran

SUMMARY:
The purpose of this study is to determine whether a top-down treatment approach, prescribing infliximab (IFX) and azathioprine (AZA) at diagnose, yields better outcome in comparison to the usual step-up treatment approach, starting with prednison and AZA or exclusive enteral nutrition (EEN) and AZA, in moderate-to-severe pediatric Crohn's disease (CD) patients.

DETAILED DESCRIPTION:
Objective: The purpose of this study is to determine whether a top-down treatment approach, prescribing IFX and AZA at diagnose, yields better outcome in comparison to the usual step-up treatment approach, starting with prednison and AZA or EEN and AZA, in moderate-to-severe pediatric CD patients.

Sample size: We will include 100 (2 x 50) patients. With these numbers a difference of 60% and 85% (= 25) can be shown at a power of 80% (2-sided α 0.05).

Study design: an international open-label randomised controlled trial Study population: Children (age 3-17 yrs) with new-onset, untreated, CD with moderate-to-severe disease activity (weighted Pediatric CD Index [wPCDAI] >40) Intervention: Patients will be randomised to either top-down or conventional step-up treatment.

Treatment arm 1: Top-down IFX treatment will consist of a total of 5 IFX infusions of 5 mg/kg (IFX induction at week 0, 2 and 6, followed by 2 maintenance infusions every 8 weeks) combined with oral AZA 2-3 mg/kg once daily. AZA therapy will continue after the last IFX infusion to maintain remission.

Treatment arm 2: Step-up treatment will consist of standard induction treatment by either oral prednisolone 1 mg/kg (maximum 40 mg) once daily for 4 weeks, followed by tapering in 6 weeks until stop, or EEN with polymeric feeding for 6-8 weeks after which normal foods are gradually reintroduced within 2-3 weeks. Either of these induction treatments will be combined with oral AZA 2-3 mg, once daily, as maintenance treatment.

Main study parameters/endpoints: Clinical remission at 52 weeks without need for additional CD related therapy or surgery. Secondary endpoints include clinical response, remission and mucosal healing at week 10 and 52, growth, quality of life and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Children (age 3-17 years, both male and female, weight >10kg) with new-onset,
* untreated CD with moderate-to-severe disease activity assessed by a wPCDAI >40 will be eligible for inclusion after a diagnosis of CD was made based on the Porto criteria

Exclusion Criteria:

Patients with the following characteristics will be excluded:

* immediate need for surgery,
* symptomatic stenosis or stricture in the bowel due to scarring,
* active perianal fistulas,
* severe co-morbidity,
* severe infection such as sepsis or opportunistic infections,
* positive stool culture,
* positive Clostridium difficile assay,
* positive tuberculin test or a chest radiograph consistent with tuberculosis or malignancy,
* those already started with CD specific therapy,
* patients with a suspected or
* definitive pregnancy

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2024-01 (Actual)

PRIMARY OUTCOMES:
Clinical remission without need for additional CD related therapy or surgery | 52 weeks
  Clinical remission is defined as a weighted Pediatric Crohn's Disease Activity Index (wPCDAI) score of less than 12.5 points

SECONDARY OUTCOMES:
Clinical response rates | 10 weeks
  Response is defined by a decrease in wPCDAI score above 17.5 points compared to baseline
Clinical remission rates | 10 and 52 weeks
  Remission is wPCDAI<12.5
Mucosal healing | 10 and 52 weeks
  Assessed by endoscopy (SES-CD) and/or fecal calprotectin (<100microgram/gram)
Change in height Z-scores | 10 and 52 weeks
Change in BMI Z-scores | 10 and 52 weeks
Change bone age | 10 and 52 weeks
Change in Tanner stage | 10 and 52 weeks
Therapy failure rates over time | 52 weeks
  Therapy failure: primary non-response, loss of response according to wPCDAI and medication intolerance
Adverse events rates | 52 weeks, and 260 weeks
  Adverse events includes therapy side effects, disease complications (fistulas, abscesses, strictures, surgery, extra-intestinal manifestations)
Cumulative therapy use | 52 weeks, and 260 weeks
Long-term yearly remission rates without need for additional CD related therapy or surgery | 260 weeks
  Clinical remission is defined as a weighted Pediatric Crohn's Disease Activity Index (wPCDAI) score of less than 12.5 points
Long-term yearly number of flares | 260 weeks
Long-term yearly clinical remission rates | 260 weeks
  Clinical remission is defined as a weighted Pediatric Crohn's Disease Activity Index (wPCDAI) score of less than 12.5 points
Long-term yearly mucosal healing (calprotectin) rates | 260 weeks
  fecal calprotectin <100microgram/gram

CONTACTS AND LOCATIONS:
Overall Officials: Lissy de Ridder, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (13):
- Belgium (2):
  - University Hospital Brussels, Brussels
  - University Hospitals Leuven, Leuven
- Helsinki University Central Hospital, Helsinki, Finland
- Netherlands (10):
  - Erasmus Medical Center, Rotterdam, South Holland
  - Academic Medical Center, Amsterdam
  - VU University Medical Center, Amsterdam
  - Amphia Hospital, Breda
  - Medisch Spectrum Twente, Enschede
  - Leiden University Medical Center, Leiden
  - Radboud University Medical Center, Nijmegen
  - Maasstad Hospital, Rotterdam
  - University Medical Center Utrecht, Utrecht
  - Isala hospital, Zwolle

REFERENCES:
- [Derived] Vuijk SA, Jongsma MME, Hoeven BM, Cozijnsen MA, van Pieterson M, de Meij TGJ, Norbruis OF, Groeneweg M, Wolters VM, van Wering H, Hummel T, Stapelbroek J, van der Feen C, van Rheenen PF, van Wijk MP, Teklenburg S, Rizopoulos D, Poley MJ, Escher JC, de Ridder L. Randomised clinical trial: First-line infliximab biosimilar is cost-effective compared to conventional treatment in paediatric Crohn's disease. Aliment Pharmacol Ther. 2024 Jun;59(12):1510-1520. doi: 10.1111/apt.18000. Epub 2024 Apr 21. PMID 38644588
- [Derived] Jongsma MME, Costes LMM, Tindemans I, Cozijnsen MA, Raatgreep RHC, van Pieterson M, Li Y, Escher JC, de Ridder L, Samsom JN. Serum Immune Profiling in Paediatric Crohn's Disease Demonstrates Stronger Immune Modulation With First-Line Infliximab Than Conventional Therapy and Pre-Treatment Profiles Predict Clinical Response to Both Treatments. J Crohns Colitis. 2023 Aug 21;17(8):1262-1277. doi: 10.1093/ecco-jcc/jjad049. PMID 36934327
- [Derived] Jongsma MME, Aardoom MA, Cozijnsen MA, van Pieterson M, de Meij T, Groeneweg M, Norbruis OF, Wolters VM, van Wering HM, Hojsak I, Kolho KL, Hummel T, Stapelbroek J, van der Feen C, van Rheenen PF, van Wijk MP, Teklenburg-Roord STA, Schreurs MWJ, Rizopoulos D, Doukas M, Escher JC, Samsom JN, de Ridder L. First-line treatment with infliximab versus conventional treatment in children with newly diagnosed moderate-to-severe Crohn's disease: an open-label multicentre randomised controlled trial. Gut. 2022 Jan;71(1):34-42. doi: 10.1136/gutjnl-2020-322339. Epub 2020 Dec 31. PMID 33384335
- [Derived] Cozijnsen MA, van Pieterson M, Samsom JN, Escher JC, de Ridder L. Top-down Infliximab Study in Kids with Crohn's disease (TISKids): an international multicentre randomised controlled trial. BMJ Open Gastroenterol. 2016 Dec 22;3(1):e000123. doi: 10.1136/bmjgast-2016-000123. eCollection 2016. PMID 28090335